CLINICAL TRIAL: NCT02608099
Title: Apixaban Evaluation of Interrupted Or Uninterrupted Anticoagulation for Ablation of Atrial Fibrillation
Acronym: AEIOU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV185-373
Record Dates: First submitted 2015-11-09; First posted 2015-11-18 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Non-valvular atrial fibrillation; Catheter ablation; Apixaban; Warfarin; Harvard Clinical Research Institute
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interrupted apixaban (Active Comparator): Apixaban dose is administered on the evening prior to the procedure; apixaban dose is held on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  Interventions: Drug: Interrupted apixaban
- Uninterrupted apixaban (Experimental): Apixaban dose is administered on the evening prior to the procedure; apixaban dose is administered on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  Interventions: Drug: Uninterrupted apixaban

INTERVENTIONS:
Drug: Interrupted apixaban — Apixaban dose is administered on the evening prior to the procedure; apixaban dose is held on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  Other Names: Interrupted Eliquis
  Arms: Interrupted apixaban
Drug: Uninterrupted apixaban — Intervention description: Apixaban dose is administered on the evening prior to the procedure; apixaban dose is administered on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  Other Names: Uninterrupted Eliquis
  Arms: Uninterrupted apixaban

SUMMARY:
The purpose of the prospective, randomized cohort in this study is to assess the safety and efficacy of 2 apixaban treatment strategies (uninterrupted versus interrupted) in subjects planned to undergo catheter ablation for the treatment of non-valvular atrial fibrillation (NVAF).

Simultaneously, a retrospective cohort of 300 warfarin-treated individuals, identified by chart review, who are matched to the prospective randomized subjects, will be identified. The purpose of the retrospective warfarin cohort is to compare the efficacy and safety of warfarin(the current clinical practice) to that of apixaban (uninterrupted, interrupted, combined uninterrupted and interrupted).

DETAILED DESCRIPTION:
Prospective, Randomized Cohort

Subjects undergoing ablation for NVAF who meet all eligibility criteria and sign informed consent will be enrolled into the study. Subjects will be treated with apixaban for ≥21 days prior to the ablation procedure (for subjects already on apixaban for ≥21 days, it is not necessary to wait 21 days before the ablation procedure. Apixaban dose will be 5 mg b.i.d. per product label, or 2.5 mg b.i.d. in subjects with 2 or more of the following: age ≥80 years, body weight ≤60 kg, or serum creatinine ≥1.5 mg/dL.

Eligible subjects will then be randomized in a 1:1 ratio to 2 peri-procedural treatment strategies:

* Uninterrupted treatment: administer the evening apixaban dose on the day prior to the procedure; administer the morning apixaban dose on the day of the procedure; administer heparin bolus before transseptal puncture to maintain a target activated clotting time [ACT] > 300 seconds; administer the evening apixaban dose after the procedure if there were no peri-procedural complications that necessitate withholding anticoagulation for longer duration.
* Interrupted treatment: administer the evening apixaban dose on the day prior to the procedure; do not administer the morning apixaban dose on the day of the procedure; administer heparin bolus before transseptal puncture to maintain a target ACT > 300 seconds; administer the evening apixaban dose after the procedure if there were no peri-procedural complications that necessitate withholding anticoagulation for longer duration.

Randomization will take place prior to the procedure (on the day of the procedure or up to 3 days prior to the procedure) and will be stratified by site.

It is anticipated that up to 360 subjects may be enrolled in order to evaluate a total of 300 randomized subjects (150 subjects per treatment arm):

Randomized subjects will continue treatment with apixaban for 1 month post procedure.

Retrospective, Warfarin Cohort In addition, a chart review of 300 warfarin-treated patients who underwent catheter ablation for NVAF on or after September 1, 2013 in the enrolling centers and who have documented follow-up in the medical record for ≥ 30 days post-ablation procedure will be performed. Patient records for warfarin-treated individuals who meet the applicable inclusion/exclusion criteria and who are matched 1:1 to a subject in the prospective, randomized cohort for age (+/- 5 years), gender and atrial fibrillation (AF) type (paroxysmal vs. persistent), will be identified. Sites will document key demographic and outcome variables. This review will be performed in a blinded manner such that site personnel are blinded to the outcome of each retrospective subject during the subject selection process. Only pre-existing data will be collected for the analysis of this cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. >18 years of age.
3. NVAF with planned catheter ablation treatment.
4. Planned anticoagulant treatment for at least 1 month after the index procedure.
5. Subject agrees to all required follow-up procedures and visits.
6. For women of childbearing potential (WOCBP):

   * Must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug.
   * Must not be breastfeeding
   * Must agree to follow instructions for method(s) of contraception for a total of 33 days post-treatment completion.
7. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a total of 93 days post-treatment completion.
8. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as described in this section.

Exclusion Criteria:

1. History of significant bleeding diathesis or coagulopathy or inability to accept blood transfusions.
2. Known hypersensitivity or contraindication to heparin or apixaban.
3. Subjects with mechanical prosthetic heart valves.
4. History of cerebrovascular accident or transient ischemic attach (TIA) within the last 6 months.
5. Prior intracranial hemorrhage.
6. End-stage renal failure (creatinine clearance rate <15 mL/minute or on dialysis treatment).
7. Hepatic disease associated with coagulopathy.
8. Current or expected systemic treatment with strong dual inducers of CYP3A4 and P-glycoprotein (e.g., rifampin, carbamazepine, phenytoin, St. John's Wort).
9. Current or expected systemic treatment with dual antiplatelet therapy, other anticoagulants, or fibrinolytics.
10. Planned or expected surgery, or other invasive procedure that would require interruption of anticoagulation within 1 month of the catheter ablation procedure.
11. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
12. Co-morbid condition(s) that could limit the subject's ability to participate in the trial or to comply with follow-up requirements, or that could impact the scientific integrity of the trial.
13. Platelet count ≤100,000/mm3.
14. Hemoglobin level <9 g/dL.
15. Any active bleeding.
16. Prisoners or subjects who are involuntarily incarcerated.
17. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Reynolds, MD, MSc, Principal Investigator — Lahey Hospital & Medical Center; Christopher P Cannon, MD, Principal Investigator — Harvard Clinical Research Organization and Cardiovascular Division Brigham and Women's Hospital
Locations (19):
- United States (19):
  - Site 0020, Huntsville, Alabama
  - Site 0005, Mission Viejo, California
  - Site 0012, New Haven, Connecticut
  - Site 0011, Trumbull, Connecticut
  - Site 0016, Pensacola, Florida
  - Site 0014, West Des Moines, Iowa
  - Site 0018, Bangor, Maine
  - Site 0004, Scarborough, Maine
  - Site 0008, Boston, Massachusetts
  - Site 0001, Burlington, Massachusetts
  - Site 0006, Kansas City, Missouri
  - Site 0021, Omaha, Nebraska
  - Site 0019, Albuquerque, New Mexico
  - Site 0002, Toledo, Ohio
  - Site 0007, Oklahoma City, Oklahoma
  - Site 0009, Philadelphia, Pennsylvania
  - Site 0010, Charleston, South Carolina
  - Site 0017, Austin, Texas
  - Site 0003, Richmond, Virginia

REFERENCES:
- [Derived] Bawazeer GA, Alkofide HA, Alsharafi AA, Babakr NO, Altorkistani AM, Kashour TS, Miligkos M, AlFaleh KM, Al-Ansary LA. Interrupted versus uninterrupted anticoagulation therapy for catheter ablation in adults with arrhythmias. Cochrane Database Syst Rev. 2021 Oct 21;10(10):CD013504. doi: 10.1002/14651858.CD013504.pub2. PMID 34674223
- [Derived] Reynolds MR, Allison JS, Natale A, Weisberg IL, Ellenbogen KA, Richards M, Hsieh WH, Sutherland J, Cannon CP. A Prospective Randomized Trial of Apixaban Dosing During Atrial Fibrillation Ablation: The AEIOU Trial. JACC Clin Electrophysiol. 2018 May;4(5):580-588. doi: 10.1016/j.jacep.2017.11.005. Epub 2017 Dec 20. PMID 29798783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Started (This number represents the intention-to-treat population.) | 148 | 152
Safety (This number represents the safety population (analyzed under the actual treatment received).) | 149 | 151
Completed (This represents the evaluable population (analyzed under assigned/randomized treatment).) | 145 | 150
Not Completed | 3 | 2
Not completed — Ablation procedure not initiated | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban | Total
Number analyzed (Participants) | 145 | 150 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (10.3) | 62.8 (9.9) | 63.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 97 | 101 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 280 patients were evaluated for ethnicity measurement.
  Participants
    number analyzed (Participants) | 135 | 145 | 280
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 134 | 143 | 277
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 283 patients were evaluated for race measurement.
  Participants
    number analyzed (Participants) | 139 | 144 | 283
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 2 | 6
    White | 133 | 141 | 274
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.46 (5.607) | 30.58 (6.441) | 30.52 (6.036)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinically-Significant Bleeding
Description: Clinically significant bleeding was defined as bleeding meeting Bleeding Academic Research Consortium (BARC) criteria type 2 or higher.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 14 | 17

2. Primary Outcome: Number of Patients With Thrombotic Events
Description: Thrombotic events were defined as a composite of non-hemorrhagic stroke and systemic thromboembolic events.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 0 | 0

3. Secondary Outcome: Number of Patients With Composite of Major Bleeding and Thrombotic Events
Description: Major bleeding was defined as bleeding meeting BARC criteria type 3 or higher. Thrombotic events were defined as a composite of non-hemorrhagic stroke and systemic thromboembolic events.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 3 | 2

4. Secondary Outcome: Number of Patients With Composite of Clinically Significant Bleeding and Thrombotic Events
Description: Thrombotic events were defined as a composite of non-hemorrhagic stroke and systemic thromboembolic events.
  Clinically significant bleeding was defined as bleeding meeting Bleeding Academic Research Consortium (BARC) criteria type 2 or higher.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 14 | 17

5. Other Pre Specified Outcome: Number of Patients With Clinically-Significant Bleeding
Description: as for outcome 1
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 17 | 17

6. Other Pre Specified Outcome: Number of Patients With Major Bleeding
Description: Major bleeding was defined as bleeding meeting BARC criteria type 3 or higher.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 3 | 2

7. Other Pre Specified Outcome: Number of Patients With Major Bleeding
Description: Major bleeding was defined as bleeding meeting BARC criteria type 3 or higher.
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 3 | 2

8. Other Pre Specified Outcome: Number of Patients With Thrombotic Events
Description: Thrombotic events were defined as a composite of non-hemorrhagic stroke and systemic thromboembolic events.
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 0 | 0

9. Other Pre Specified Outcome: Number of Patients With Composite of Clinically Significant Bleeding and Thrombotic Events
Description: as for outcome 4
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 14 | 17

10. Other Pre Specified Outcome: Number of Patients With Composite of Major Bleeding and Thrombotic Events
Description: Thrombotic events are defined as a composite of non-hemorrhagic stroke and systemic thromboembolic events.
  Major bleeding is defined as bleeding meeting BARC criteria type 3 or higher.
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 3 | 2

11. Other Pre Specified Outcome: Number of Patients With TIAs or Non-Hemorrhagic Strokes
Description: Number of Patients who had TIAs or non-hemorrhagic strokes.
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 1 | 1

12. Other Pre Specified Outcome: Number of Patients With TIAs or Non-Hemorrhagic Strokes
Description: This measurement includes TIAs or non-hemorrhagic strokes.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 1 | 1

13. Other Pre Specified Outcome: Number of Patients With Death
Description: Death is included in this measurement.
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 0 | 0

14. Other Pre Specified Outcome: Number of Patients With Cardiovascular Death
Description: Cardiovascular death is included in this measurement.
Time Frame: Enrollment to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 0 | 0

15. Other Pre Specified Outcome: Number of Patients With Death
Description: Death is included in this measurement.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 0 | 0

16. Other Pre Specified Outcome: Number of Patients With Cardiovascular Death
Description: Cardiovascular death is included in this measurement.
Time Frame: Randomization to 1 month post catheter ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
Number analyzed (Participants) | 145 | 150
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Month
Description: Treatment Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term. The safety population was used to report the SAEs and AEs.
Groups:
- Interrupted Apixaban: Apixaban dose is administered on the evening prior to the procedure; apixaban dose is held on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  Interrupted apixaban: Apixaban dose is administered on the evening prior to the procedure; apixaban dose is held on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  A total of 149 patients were included in the "Interrupted Apixaban" arm from the safety population (patients were analyzed under the actual treatment received).
- Uninterrupted Apixaban: Apixaban dose is administered on the evening prior to the procedure; apixaban dose is administered on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  Uninterrupted apixaban: Intervention description: Apixaban dose is administered on the evening prior to the procedure; apixaban dose is administered on the morning of the procedure; apixaban dose is administered on the evening after the procedure if there were no peri-procedural complications that necessitated withholding anticoagulation for longer duration.
  A total of 151 patients were included in the "Uninterrupted Apixaban" arm from the safety population (patients were analyzed under the actual treatment received).
Arm/Group | Interrupted Apixaban | Uninterrupted Apixaban
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/151
Serious Adverse Events (participants affected / at risk) | 14/149 | 15/151
Other Adverse Events (participants affected / at risk) | 72/149 | 75/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interrupted Apixaban (N=149) | Uninterrupted Apixaban (N=151)
Arrhythmia Supraventricular (Cardiac disorders) | 2 | 1
Blindness Transient (Eye disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Catheter Site Haemorrhage (General disorders) | 1 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 2 | 3
Atrial Flutter (Cardiac disorders) | 2 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiac Perforation (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 1
Sinus Arrest (Cardiac disorders) | 1 | 0
Catheter Site Pain (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interrupted Apixaban (N=149) | Uninterrupted Apixaban (N=151)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 1
Arrhythmia supraventricular (Cardiac disorders) | 10 | 9
Atrial fibrillation (Cardiac disorders) | 13 | 7
Atrial flutter (Cardiac disorders) | 7 | 3
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 3
Pericarditis (Cardiac disorders) | 1 | 2
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Blindness transient (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 7
Catheter site bruise (General disorders) | 3 | 3
Catheter site discharge (General disorders) | 2 | 3
Catheter site haematoma (General disorders) | 5 | 2
Catheter site haemorrhage (General disorders) | 8 | 5
Catheter site pain (General disorders) | 7 | 3
Catheter site swelling (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Infusion site pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 6 | 6
Oedema peripheral (General disorders) | 2 | 5
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 3
Fluid retention (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 3 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT02608099/SAP_000.pdf
  • Study Protocol (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT02608099/Prot_001.pdf